CLINICAL TRIAL: NCT03021668
Title: A Randomized Control Trial of Prevena Peel & Place Dressing Versus Standard Closure for Patients Undergoing Pancreaticoduodenectomy Who Have Undergone Neoadjuvant Chemotherapy or Biliary Stent Placement
Brief Title: Comparison Between Wound Vacuum Dressing and Standard Closure to Reduce Rates of Surgical Site Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00109564
Record Dates: First submitted 2017-01-06; First posted 2017-01-16 (Estimated); Results first posted 2019-02-12 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Surgical Site Infection; Pancreatic Neoplasms; Pancreatic Cancer; Chemotherapy Effects; Chemoradiation; Surgical Wound; Wound Complication
MeSH Terms: conditions — Surgical Wound Infection; Pancreatic Neoplasms; Surgical Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prevena Peel & Place Dressing for wound closure (Experimental): In the participants randomized to this arm the surgical site will be closed using Prevena Peel & Place Dressing.
  Interventions: Device: Prevena Peel & Place Dressing
- Standard closure of the wound (Placebo Comparator): In the participants randomized to this arm the surgical site will be closed using the standard closure technique.
  Interventions: Other: Standard Closure of the Surgical Incision

INTERVENTIONS:
Device: Prevena Peel & Place Dressing — Prevena Peel & Place Dressing is a device that can be used for closure of the surgical site. It provides negative pressure to the surgical wound
  Arms: Prevena Peel & Place Dressing for wound closure
Other: Standard Closure of the Surgical Incision — This would involve standard closure of the incision site
  Arms: Standard closure of the wound

SUMMARY:
Pancreaticoduodenectomy is associated with high perioperative morbidity, with surgical site infection (SSIs) being one of the most common complications. A retrospective study at Hopkins on SSIs in these patients identified the rate of SSIs to be 16.7% and pre-operative bile stent/drain and neoadjuvant chemotherapy were independent predictors of surgical site infection. Patients with these factors having a predicted risk of up to 32%. Another subsequent retrospective study demonstrated that the use of negative pressure wound therapy device was significantly associated with a decrease in the rate of SSIs.

The hypothesis of the investigator(s) for the current study is that placement of Prevena Peel & Place Dressing (Negative Pressure Wound Therapy, NPWT) in patients undergoing pancreaticoduodenectomy who are at high risk of SSIs will result in a significant decrease in their SSI rate.

DETAILED DESCRIPTION:
Although outcomes of pancreaticoduodenectomy have improved, it remains a procedure with a high perioperative complication rate. Surgical site infection is one of the most common complications after pancreaticoduodenectomy. In a retrospective review of all patients who underwent pancreaticoduodenectomy at Johns Hopkins between 9/2011 and 8/2014, a total of 679 patients, 30-day surgical site infection was observed in 16.7%. By univariate analysis, perioperative blood transfusion, operative time greater than 7 hours, preoperative chemotherapy and/or radiation, bile stent, absence of a superficial wound vacuum closure device, and vascular resection were associated with surgical site infection (all, p<0.05). On multivariable analysis, pre-operative bile stent/drain and neoadjuvant chemotherapy were independent predictors of surgical site infection (all, p<0.001). Studies in colorectal patients have found an estimated cost of up to $1400 per patient secondary to prolonged hospitalization, wound care, and wound complications in patients with procedures complicated by a surgical site infection. Furthermore, in another study of 1144 patients undergoing pancreaticoduodenectomy between 1995 and 2011 at Johns Hopkins Hospital, post-operative complications delayed time to adjuvant therapy, decreased median survival.

The hypothesis of the investigator(s) is that placement of Prevena Peel & Place Dressing using the standard Acelity vacuum dressing after suture on patients undergoing pancreaticoduodenectomy at highest risk of infection will result in a significant decrease in surgical site infection rate. The investigator(s) plan to perform a randomized control trial where the patients who have had pre-operative bile stent/drain placement and/or neoadjuvant chemotherapy will undergo closure with Prevena Peel & Place Dressing using the standard Acelity vacuum dressing after suture versus standard closure. The investigator(s) will then follow the participant(s) for 30 days postoperatively to determine surgical site infection and other perioperative complication rate.

ELIGIBILITY:
Inclusion Criteria:

* Patient to undergo pancreaticoduodenectomy for pancreatic tumors at the Johns Hopkins Hospital
* Patient treated with neoadjuvant chemotherapy with or without radiation therapy prior to surgical resection, AND/OR placement of a biliary stent and/or drain for biliary tree decompression

Exclusion Criteria:

* Age 18 years or younger
* Laparoscopic or robotic pancreaticoduodenectomy
* Patient did not undergo either placement of a preoperative biliary stent/drain or neoadjuvant chemotherapy with or without radiation therapy
* All patients who are have known allergies or are sensitive to silver and acrylic adhesives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Weiss, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prevena Peel & Place Dressing for Wound Closure | Standard Closure of the Wound
Started | 62 | 62
Completed | 62 | 61
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prevena Peel & Place Dressing for Wound Closure | Standard Closure of the Wound | Total
Number analyzed (Participants) | 62 | 61 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (9.3) | 66.1 (9.0) | 66.2 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 27 | 58
  Male | 31 | 34 | 65
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 8 | 12
  White | 55 | 47 | 102
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 6 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 62 | 61 | 123
Neoadjuvant therapy [Count of Participants; unit: Participants] | 44 | 33 | 77
American Society of Anesthesiologists (ASA) class [Count of Participants; unit: Participants] — The patients were graded according to the American Society of Anesthesiologists risk scoring system. Patients are scores between I and IV based on their operative risk.
  ASA I: A normal healthy patient. ASA II: A patient with a mild systemic disease. ASA III: A patient with a severe systemic disease that is not life-threatening. ASA IV: A patient with a severe systemic disease that is a constant threat to life.
  Participants
    ASA I/II | 11 | 14 | 25
    ASA III/IV | 51 | 47 | 98
Preincisional prophylactic antibiotic [Count of Participants; unit: Participants] | 62 | 61 | 123
Preoperative biliary stenting [Count of Participants; unit: Participants] | 51 | 51 | 102

OUTCOME MEASURES:

1. Primary Outcome: Rate of Surgical Site Infection
Description: Surgical site infection will be diagnosed and classified based on the World Health Organization definition into superficial Infection (involving only skin and subcutaneous tissue of incision), deep incisional (involving deep tissues) or organ/space (involving organs and spaces other than the incision which was opened or manipulated during operation)
Time Frame: Within 30 days of the operation
Measure: Count of Participants; unit: Participants
Arm/Group | Prevena Peel & Place Dressing for Wound Closure | Standard Closure of the Wound
Number analyzed (Participants) | 62 | 61
Participants | 6 | 19
Statistical Analysis 1: Comparison: Prevena Peel & Place Dressing for Wound Closure vs Standard Closure of the Wound; Test type: Equivalence — Chi2 test was performed to analyze difference in rates of Surgical Site Infections (SSIs) between the two groups; p = 0.003, Chi-squared

2. Secondary Outcome: Prolonged Length of Stay, Measured in Days
Description: Length of stay of patient at the hospital from date of surgery
Time Frame: Within 10 days of surgery
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Prevena Peel & Place Dressing for Wound Closure | Standard Closure of the Wound
Number analyzed (Participants) | 62 | 61
days | 7 [7 to 10] | 8 [7 to 10]
Statistical Analysis 1: Comparison: Prevena Peel & Place Dressing for Wound Closure vs Standard Closure of the Wound; Test type: Equivalence — Students' T-test was used to evaluate any difference in length of stay between the two groups; p = 0.23, t-test, 2 sided

3. Secondary Outcome: Rate of Readmission for Surgical Site Infections (SSIs)
Description: Any readmission for surgical site infections (SSIs) related to the surgery within the first 30 days after surgery
Time Frame: Within 30 days of operation
Measure: Count of Participants; unit: Participants
Arm/Group | Prevena Peel & Place Dressing for Wound Closure | Standard Closure of the Wound
Number analyzed (Participants) | 62 | 61
Participants | 3 | 6

4. Secondary Outcome: 30-d Readmission
Description: Need for 30-day readmission
Time Frame: Within 30 days of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Prevena Peel & Place Dressing for Wound Closure | Standard Closure of the Wound
Number analyzed (Participants) | 62 | 61
Participants | 5 | 12

ADVERSE EVENTS:
Time Frame: Within 90 days of surgery
Arm/Group | Prevena Peel & Place Dressing for Wound Closure | Standard Closure of the Wound
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/61
Other Adverse Events (participants affected / at risk) | 7/62 | 15/61
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prevena Peel & Place Dressing for Wound Closure (N=62) | Standard Closure of the Wound (N=61)
Postoperative pancreatic fistula (Hepatobiliary disorders) | 3 (3) | 7 (7)
Delayed gastric emptying (Gastrointestinal disorders) | 6 (6) | 6 (6) — Postoperative delayed gastric emptying
Postoperative respiratory complications (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 8 (8)

LIMITATIONS AND CAVEATS:
The study was conducted at a high volume center for pancreatic surgery with a broad experience using Negative-Pressure Wound Therapy (NPWT), and therefore there is a question about the generalizability of the reductions we observed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/68/NCT03021668/Prot_SAP_000.pdf